CLINICAL TRIAL: NCT00920036
Title: Adjunctive Biofeedback Intervention for OIF-OEF PTSD
Brief Title: Adjunctive Biofeedback Intervention for Operation Iraqi Freedom/Operation Enduring Freedom (OIF-OEF) Post Traumatic Stress Disorder (PTSD)
Acronym: ABIOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Arkansas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 203987
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Post-traumatic Stress Disorder
Keywords: PTSD; Combat; Biofeedback; Psychophysiology
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Eight subjects were trained to utilize a handheld biofeedback device
  Interventions: Device: StressEraser
- Arm 2 (No Intervention): usual care

INTERVENTIONS:
Device: StressEraser — A hand-held biofeedback device that facilitates resonant frequency of respiration
  Arms: Arm 1

SUMMARY:
Objective:

The aims are to examine the feasibility and acceptability of a handheld biofeedback device as an adjunct treatment for Post Traumatic Stress Disorder (PTSD) and to estimate its clinical effect size. A recent summary of 22 studies on OIF/OEF (Operation Iraqi Freedom/Operation Enduring Freedom) veterans revealed that many individual and system factors (e.g., stigma, concern about promotion/employment, lack of providers) prevented access to mental health services. For veterans who did seek help, the largest treatment trials of pharmacologic, outpatient psychotherapy, and residential treatment programs were not very effective. Currently, prolonged exposure therapy is the most validated PTSD treatment. The VHA enrollees from OIF/OEF are more likely to live in rural areas, hindering them from pursuing treatment due to travel distance and time commitment. Thus, new treatments and delivery methods are urgently needed.

A substantial body of preclinical literature documents autonomic nervous system (ANS) dysregulation in patients with PTSD. Preliminary results suggest that portable heart rate variability (HRV)/respiratory sinus arrhythmia (RSA) biofeedback is a promising adjunct treatment for autonomic arousal disorders. The StressEraser, a HRV/RSA biofeedback device, is indicated for relaxation, relaxation training, and stress reduction. This small handheld device measures and displays real-time RSA via an infrared finger sensor.

Research Plan:

The investigators were able to randomize 16 OIF/OEF veterans receiving care for PTSD at CAVHS community-based outpatient clinics (CBOCs) to a 24-week course of StressEraser use (N=8) versus usual care (N=8). A trouble-shooting phone call to participants occurred at 6 weeks. Follow-up clinical assessments occurred at 12 and 24 weeks.

Methods:

The baseline assessment consisted of a screening interview for comorbid anxiety and substance use disorders, the Clinician Administered PTSD Scale (CAPS), the 9-item depression Patient Health Questionnaire (PHQ-9), and a quality of life measure (Quality of Well-Being Scale-Self Administered [QWB-SA]). In addition, psychophysiologic assessment of reactivity and attentional bias to combat-related PTSD relevant stimuli occurred through virtual reality (VR) and acoustic startle stimuli at the North Little Rock psychophysiologic reactivity lab. The StressEraser group was trained to operate the device at baseline and instructed to use it for 5-20 minutes daily before bedtime for 24 weeks.

At six weeks, a research assistant phoned the StressEraser group to address any problems with the device and the usual care group to insure adherence with ongoing treatment. The 12-week assessment involved phoning both groups to administer the psychometric measures (CAPS, PHQ-9, and QWB-SA). At 24 weeks, the sample returned to the lab for administration of the psychometric measures and assessment of psychophysiologic reactivity.

The subjects in the StressEraser group returned the device. The time spent using the StressEraser and the total number of resonant frequency respirations were the feasibility measures. The StressEraser logged the date, time, and duration of use and the amount of resonant frequency breathing, which is the resonance between the respiratory and baroreflex rhythms, the two primary sources of cardiac stimulation. Acceptability was measured through a short debriefing interview.

DETAILED DESCRIPTION:
The aims of this proposal are to examine the feasibility and acceptability of using a handheld biofeedback intervention as an adjunct treatment for Post Traumatic Stress Disorder (PTSD) and to estimate the effect size of the biofeedback intervention as an adjunct treatment for PTSD.

A recent RAND Corporation Report summarized 22 studies of OIF/OEF (Operation Iraqi Freedom/Operation Enduring Freedom) veterans, giving a typical range of 5-15% for veterans meeting diagnostic criteria for PTSD, with some studies reporting rates as high as 30%. Of those active duty service members meeting criteria for mental health referral based on the post-deployment health assessment, only about half (41.8-61.0%) received mental health services. Many individual and system factors (e.g., stigma, concern about promotion/employment, wait times, lack of providers) prevented access.

Historically, for those veterans who access treatment for combat-related PTSD, the largest treatment trials of pharmacologic, outpatient psychotherapy, and residential treatment programs have not shown these treatments to be very effective. More recently, the Institute of Medicine has recommended prolonged exposure therapy as the most validated of PTSD treatments. However, rural OIF/OEF veterans are hindered by travel distance and the time commitment necessary to receive such recommended treatments. The VA Office of Rural Health reported that VHA enrollees from OIF/OEF were more likely to live in rural areas. Thus, new treatments and new treatment delivery methods are urgently needed.

A substantial historic and growing preclinical literature documents autonomic nervous system (ANS) dysregulation in patients with PTSD. Preliminary results suggest that portable heart rate variability (HRV)/ respiratory sinus arrhythmia (RSA) biofeedback appears to be a promising adjunct treatment for disorders of autonomic arousal. The StressEraser, a HRV/RSA biofeedback device, is indicated for relaxation, relaxation training, and stress reduction. The StressEraser is a small handheld device that measures and displays real-time RSA, a measure of HRV, via an infrared finger sensor.

We will randomize 30 OIF/OEF veterans receiving care for PTSD at CAVHS community-based outpatient clinics (CBOC's) to a 24-week course of StressEraser use (N=15) versus usual care (N=15). The baseline assessment will consist of a screening interview for comorbid anxiety and substance use disorders, the Clinician Administered PTSD Scale (CAPS), the 9-item depression Patient Health Questionnaire (PHQ-9) to determine symptoms of depression, and a quality of life measure (Quality of Well-Being Scale-Self Administered [QWB-SA]).

In addition, subjects will participate in assessment of psychophysiologic measures in response to virtual reality (VR) and acoustic startle stimuli and attentional bias measures to combat-related PTSD relevant stimuli. Subjects in the StressEraser group will be trained to use and demonstrate proficiency in using the device at completion of the baseline assessment. These subjects will be instructed to use the StressEraser for 5-20 minutes daily before bedtime for 24 weeks. Follow-up assessments will occur at 12 and 24 weeks after baseline for both the StressEraser and usual care subjects. Subjects will be contacted by phone at 6 weeks to address any problems using the StressEraser (intervention group) and to insure adherence with ongoing treatment in the usual care group. The 12-week assessments will occur over the phone and address current symptom severity of PTSD (CAPS) and depression (PHQ-9) and health-related quality of life with the QWB-SA. The 24-week assessment will be in-person at the psychophysiologic reactivity lab in North Little Rock for repeat assessment of psychophysiologic measures through VR and acoustic startle stimuli and attentional bias measures to combat-related PTSD relevant stimuli and will include the psychometric measures. The subject will be asked to bring the StressEraser with him/her to the 24-week assessment to document the duration and frequency of use.

Feasibility will be measured by the amount of time the subject spends using the StressEraser. The StressEraser logs the date, time, and duration of use. It also logs the amount of resonant frequency breathing achieved, which is the resonance between the respiratory and baroreflex rhythms, the two primary sources of cardiac stimulation. This information can be easily downloaded from the StressEraser device. The feasibility measures will be total duration of use and total number of resonant frequency respirations.

Acceptability will be measured using a short debriefing interview at 12 weeks and a longer debriefing interview at 24 weeks. Additional measures will include change in CAPS, PHQ-9, and QWB-SA scores measured at baseline, 12, and 24 weeks and changes in psychophysiologic reactivity at 24 weeks compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* OIF/OEF veterans
* diagnosed with PTSD
* receiving mental health treatment at Community Based Outpatient Clinics or PTSD clinics in North Little Rock

Exclusion Criteria:

* diagnosis of schizophrenia
* daytime dose of benzodiazepines, beta-blockers, and stimulant medication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-02; Primary Completion 2011-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
feasibility and acceptance using qualitative measures | 6 months

SECONDARY OUTCOMES:
Clinician-Administered PTSD Scale (CAPS) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A Kimbrell, MD, Principal Investigator — Central Arkansas Veterans Healthcare System (North Little Rock)